CLINICAL TRIAL: NCT00424359
Title: A Prospective Study of Clinical Indices as Predictors of Ambulatory Effectiveness in Multiple Sclerosis
Brief Title: Ambulation Study in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Brown, Theodore R., M.D., MPH (Individual)
Responsible Party: Theodore R. Brown, MD Mph, MS Center at Evergreen
Other Study IDs: WIRB 20050607; Pfizer Inc; Independent Grants 235-14-22; NCT01355250 (obsolete NCT alias)
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Sclerosis
Keywords: Mulitple Sclerosis; Ambulation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study comparing clinical tests of walking and balance. The goal of this study is to discover which of those tests are best at predicting walking problems due to MS.

DETAILED DESCRIPTION:
This study includes:

Three study visits to the MS Center at Evergreen; wearing a pedometer for two, one-week periods to record walking during regular daily activities; keeping a diary for any walking problems such as falls and slips.

Subjects must meet the following criteria:

Diagnosis of MS (any form); 18-70 years of age; be on stable MS treatment OR no MS treatment for the last three months; no scheduled hospitalization in the next six months.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have sufficient cognitive ability to maintain a falls diary and follow instructions for wearing the pedometer
* Subject must have clinically definite MS according to McDonald criteria
* Subject must have EDSS between 0-6.5
* Subject must be aged 18-70
* Subjects must be given informed consent
* Subjects must be stable on disease modifying therapy or no therapy for at least three months before entry into study

Exclusion Criteria:

* No MS relapse within the last 30 days
* Subjects must have no scheduled major hospitalizations or surgical procedures during the study time frame. Hospitalization during the study may result in removal from the study
* Medical conditions other than MS that might significantly impact ambulatory activity (such as angina pectoris) in the judgement of the investigators
* History or suspicion of non-compliance in the judgement of the investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Multiple Sclerosis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2005-04; Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Brown, MD, MPH, Principal Investigator — MS Center at Evergreen